CLINICAL TRIAL: NCT03038425
Title: Does Continuous Adductor Canal Nerve Block Improve the Quality of Recovery for Outpatient Total Knee Arthroplasty Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20160937
Record Dates: First submitted 2017-01-20; First posted 2017-01-31 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Arthroplasty, Replacement, Knee; Nerve Block; Anesthesia, Regional; Ambulatory Surgical Procedures
MeSH Terms: interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline infusion (Placebo Comparator): Participants in this group will receive normal saline infusion (5ml/hr, patient controlled bolus 5ml, lockout 30min) in the adductor canal, starting in PACU on post-operative day 0 and continuing for 96 hours
  Interventions: Drug: Normal Saline
- Ropivacaine infusion (Active Comparator): Participants in this group will receive ropivacaine 0.2% infusion (5ml/hr, patient controlled bolus 5ml, lockout 30min) in the adductor canal, starting in PACU on post-operative day 0 and continuing for 96 hours
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Normal Saline — This is the placebo intervention - normal saline infused in the adductor canal via a catheter. There are no anticipated therapeutic effect
  Arms: Saline infusion
Drug: Ropivacaine — This is the treatment intervention - ropivacaine 0.2% infused in the adductor canal via a catheter. This will provide analgesia to the knee after TKA
  Arms: Ropivacaine infusion

SUMMARY:
This is a randomized, double-blinded pilot study to determine whether patients undergoing ambulatory total knee arthroplasty (TKA) using a subvastus approach benefit from the addition of a continuous adductor canal nerve block (cACB) catheter along with an existing multimodal approach to postoperative analgesia. Outcomes include the 15-item Quality of Recovery Scale (QoR-15) (Miles 2016), pain scores, opioid consumption, opioid-free days, functional outcome as measured by the Time Up and Go (TUG) test, patient satisfaction, patient's rating of catheter effectiveness, and complications.

ELIGIBILITY:
Inclusion Criteria:

1. patient characteristics suitable for subvastus approach as determined by single surgeon
2. patients willing to undergo ambulatory surgery
3. ability to read and verbally communicate via either English or French

Exclusion Criteria:

1. age > 80
2. driving distance greater than 1 hour from hospital
3. no willing caregiver at home on night of surgery
4. renal failure requiring dialysis
5. Insulin-dependent diabetes mellitus
6. BMI > 45
7. allergy to study medications
8. pre-existing neurologic deficit involving the ipsilateral limb
9. chronic high dose opioid use (defined as >200mg/day of morphine equivalent for over 2 weeks).
10. inability to use or manage cACB catheter and pump independently at home
11. inability or refusal to cryocompressive therapy device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery Scale 15 (QoR-15) | at 4pm on post-operative day (POD) 1
  QoR-15 is a validated scale calculated from a 15-question patient questionnaire. It is an aggregate score that evaluates recovery after surgery.

SECONDARY OUTCOMES:
Quality of Recovery Scale 15 (QoR-15) | POD 2-4 + 7
Pain score at rest | POD 1-4 + 7
  Patients will rate their pain on a scale of 0-10
Pain score with activity | POD 1-4 + 7
  Patients will rate their pain on a scale of 0-10
Tapentadol consumption | POD 1-4 + 7
  Daily tapentadol use in milligrams
Patient satisfaction | POD 1-4 + 7
  Patients will be asked "are you satisfied with your pain control"
Vital signs - blood pressure, heart rate, oxygen saturation | twice daily POD 1-4
  These measurements will be obtained via post-operative home monitoring system
Patient-rated catheter effectiveness | POD 1-4
  Patients will be asked "do you think the nerve block catheter is helpful? Rate on a 5-point scale"
Catheter specific complications | POD 1-4
  Patients will be asked daily to report these potential nerve block catheter related issues: (1) leakage around the dressing (2) occlusion/blockage of the pump (3) inadvertent catheter disconnection (4) swelling around the catheter site (5) bleeding or bruising around the catheter site (6) other complications
Peri-operative complications | POD 30
  Significant peri-operative complications resulting in return to emergency department, re-admission after discharge, or return to operating room will be reported
Timed-up-and-go (TUG) test | POD 14
  TUG is a validated test to assess a person's mobility. It has been used to evaluate functional recovery after orthopedic surgeries. This will be administered on POD 14 at the surgeon's office during the post-operative follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BY Wong, MD, Principal Investigator — The Ottawa Hospital, University of Ottawa
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided